CLINICAL TRIAL: NCT04851327
Title: Behavioural Correlates of Wasting: a Pilot Satiation Study With Children Attending a Tertiary Feeding Clinic
Brief Title: Satiation Study With Children Attending a Tertiary Feeding Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: University of Stirling (Other); University of Ghana (Other)
Responsible Party: Principal Investigator, Charlotte Wright, Professor of Community Child Health, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NHSGGC290906
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Undernutrition; Underweight
MeSH Terms: conditions — Malnutrition; Thinness

STUDY DESIGN:
Intervention Model Description: cross-over energy compensation study, participants acting as their own controls
Who Masked: Participant, Outcomes Assessor
Masking Description: Two similar tasting drinks will be used in random order, one low and one high energy After a standardised meal, the weight of food consumed will be measured by an observer blind to which supplement has been used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High energy (Experimental): Child will be given a high energy drink: a flavoured high energy milk or juice-based drink, used clinically to supplement the diet of preschool children (either Pediasure plus or Duocal). This will provide 1.5 kcals per ml in various flavours as preferred. The amount given will supply 10% of the child's daily energy requirements per Kg - for example for a 2-year-old child weighing 15 KG this would be 80 mls of drink supplying 120 Kcal.
  They will be given 10 minutes to drink the preload and 30 minutes after this they will eat lunch containing a range of pre-packaged foods of known energy content suitable for their age, chosen in consultation with the parents.
  Interventions: Behavioral: High Energy preload; Behavioral: Test meal
- Low energy (Experimental): Child will be given a low energy drink of the same volume selected to be as similar as possible to the high energy drink, made either of skim milk or sugar free fruit juice, with a similar sugar free flavour; for above example this will supply 25 kcal.
  They will be given 10 minutes to drink the preload and 30 minutes after this they will eat lunch containing the same range of pre-packaged foods as above.
  Interventions: Behavioral: Low energy preload; Behavioral: Test meal

INTERVENTIONS:
Behavioral: High Energy preload — Tests the extent to which participants reduce their intake at a meal following ingestion of a high energy preload drink
  Other Names: Satiation study
  Arms: High energy
Behavioral: Low energy preload — Tests the amount participants eat at a meal following ingestion of a low energy preload drink
  Other Names: Satiation study
  Arms: Low energy
Behavioral: Test meal — Test meal to follow low or high energy preload

SUMMARY:
This is a pilot study of children attending the Glasgow feeding clinic (GFC) which looks after children with severe feeding problems who commonly have low appetite and extreme thinness. The investigators want to find out if thin children respond to food in the same way, using an established method to assess energy compensation.

DETAILED DESCRIPTION:
Thinness occurs as a result of undereating, but it is not always clear why an individual child has not eaten enough, or how to get them to eat more. There is a need to understand the child characteristics that predispose to undereating and the how these operate, in order to design more effective treatment and prevention programmes. The Glasgow feeding clinic (GFC) looks after a range of children with severe feeding problems who commonly have low appetite and extreme thinness.

A Ghanaian student will come to Glasgow, funded by the Glasgow University /Scottish funding council Global Challenges Research fund, to learn these techniques to use in future PhD research. The student will conduct a pilot study of children attending the GFC. The student will invite 40 families to complete our standardised online questionnaire (ICFET) about their child's eating behaviour and collate existing growth measurements as well as their feeding history.

A standardised energy compensation study will then be undertaken in 20 of the thinnest children. At two visits at least a week apart, the children will be given one of two similar tasting drinks in random order, one with very few calories and another with extra, without them knowing which is which. After 30 minutes they will eat as much as they want of a standardized lunch. All foods and drinks offered will be weighed before and after, to calculate the amount of energy eaten in total after the low energy drink, compared to the high energy drink.

ELIGIBILITY:
Inclusion Criteria:

* Currently attending Glasgow Feeding Clinic or seen within the last 2 years.
* Completed ICFET questionnaire and eating solid food at least weekly.
* Body mass index < 9th centile.
* Within 40 minutes car travel from study centre

Exclusion Criteria:

* Patient or family member shielding from COVID.
* Not able to swallow safely
* Not taking solid foods
* Fully tube fed: i.e. receiving more than 75% of energy requirements from tube feeding.

No measurements

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Compensation index | Calculated on day 8, after consumption of 2nd test meal
  The difference in energy consumed after high compared to low energy preload as percent of energy in preload

SECONDARY OUTCOMES:
total energy consumed per study day | Calculated on day 8, after consumption of 2nd test meal
  The total amount of energy consumed form preload plus meal after high compared to low energy preload

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M Wright, MD, Principal Investigator — University of Glasgow
Locations (1):
- New Lister building, Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data may be made available on request